CLINICAL TRIAL: NCT04971343
Title: Evaluation of the Beckman Coulter Access HIV Ag/Ab Combo Assay as an Aid in the Diagnosis of HIV-1 and/or HIV-2 Infection: EU Clinical Trial Protocol
Brief Title: Access HIV Ag/Ab Combo Assay - European Union (EU) Clinical Trial Protocol
Acronym: HIV-EU-11-18
Status: Completed | Type: Observational
Sponsor: Beckman Coulter, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: DC-TR18-0410
Record Dates: First submitted 2021-07-12; First posted 2021-07-21 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: HIV I Infection; HIV-2 Infection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- Unselected blood donors
  Interventions: Diagnostic Test: Access HIV_blood donor; Diagnostic Test: Access HIV_Canada's requirements_Blood donor
- Hospitalized patients
  Interventions: Diagnostic Test: Access HIV_Hospitalized patient
- Known HIV-1 Ab positive
  Interventions: Diagnostic Test: Access HIV_known HIV-1 antibody positives; Diagnostic Test: Access HIV_Canada's requirements_HIV positive
- Known HIV-2 Ab positive
  Interventions: Diagnostic Test: Access HIV_known HIV-2 antibody positives; Diagnostic Test: Access HIV_Canada's requirements_HIV positive
- Known Acute HIV-1 p24 Ag positive
  Interventions: Diagnostic Test: Access HIV_known HIV-1 p24 Ag positive; Diagnostic Test: Access HIV_Canada's requirements_HIV positive; Diagnostic Test: Access HIV_Canada's requirements_P24 Positive

INTERVENTIONS:
Diagnostic Test: Access HIV_blood donor — Samples will be tested with both reference HIV Ag/Ab combo assay and Access HIV Ag/Ab combo assay according to respective IFU to determine non-reactive, initially reactive, and repeatedly reactive. Reference assay will be Roche - Cobas - Elecsys® HIV Duo .
  * All initially reactive specimen results will be tested in duplicate per IFU .
  * All RR specimens will be confirmed using testing including ImmunoBlot, Western Blot or HIV-1/HIV-2 differentiation test and HIV-1 PCR, RNA (if Immunoblot, WesternBlot or differentiation test is negative or indeterminate; if Immunoblot, WesternBlot or differentiation test is positive for HIV-2 then HIV-1 PCR will not be tested).
  Groups: Unselected blood donors
Diagnostic Test: Access HIV_Hospitalized patient — All samples will be tested with both reference HIV Ag/Ab combo assay and Access HIV Ag/Ab combo assay according to respective IFU to determine non-reactive, initially reactive, and repeatedly reactive. Reference assay will be Abbott Architect HIV Ag/Ab combo assay for hospitalized patient.
  * All initially reactive specimen results will be tested in duplicate per IFU .
  * All RR specimens will be confirmed using testing including ImmunoBlot, Western Blot or HIV-1/HIV-2 differentiation test and HIV-1 PCR, RNA (if Immunoblot, WesternBlot or differentiation test is negative or indeterminate; if Immunoblot, WesternBlot or differentiation test is positive for HIV-2 then HIV-1 PCR will not be tested).
  Groups: Hospitalized patients
Diagnostic Test: Access HIV_known HIV-1 antibody positives — Samples will be tested with both reference HIV Ag/Ab combo assay and Access HIV Ag/Ab combo assay according to respective IFU to determine non-reactive, initially reactive, and repeatedly reactive. Reference assay will be Abbott Architect HIV Ag/Ab combo assay .
  * All initially reactive specimen results will be tested in duplicate per IFU .
  * For the known positive cohorts (sensitivity cohorts), samples will be identified as positive at enrollment/time of testing according to inclusion criteria prior to testing or in parallel of testing with Access and Reference HIV Ag/Ab combo assays.
  In case of discrepant results or concordant negative results between Access and Reference HIV Ag/Ab combo assay among known HIV-1 antibody positive patients, the IB/WB test will be repeated by the site to confirm sample status. If this IB/WB result is negative or indeterminate, the sample will be excluded from the statistical analysis
  Groups: Known HIV-1 Ab positive
Diagnostic Test: Access HIV_known HIV-2 antibody positives — Samples will be tested with both reference HIV Ag/Ab combo assay and Access HIV Ag/Ab combo assay according to respective IFU to determine non-reactive, initially reactive, and repeatedly reactive. Reference assay will be Abbott Architect HIV Ag/Ab combo assay.
  * All initially reactive specimen results will be tested in duplicate per IFU .
  * For the known positive cohorts (sensitivity cohorts), samples will be identified as positive at enrollment/time of testing according to inclusion criteria prior to testing or in parallel of testing with Access and Reference HIV Ag/Ab combo assays.
  Groups: Known HIV-2 Ab positive
Diagnostic Test: Access HIV_known HIV-1 p24 Ag positive — All samples will be tested with both Reference HIV Ag/Ab combo assay and Access HIV Ag/Ab combo assay according to respective IFUs/study guide to determine non-reactive (NR), initially reactive (IR), and repeatedly reactive (RR). Reference assay will be Abbott - ARCHITECT HIV Ag/Ab Combo Assay.
  * Due to volume constraints, all known HIV-1 p24 Ag positive samples that will be tested during the EU HIV clinical trial will be tested in singulare only with the Reference HIV Ag/Ab combo assay, and in singulare and then in duplicate if IR with Access HIV Ag/Ab combo assay.
  * For the known positive cohorts (sensitivity cohorts), samples will be identified as positive at enrollment/time of testing according to inclusion criteria prior to testing or in parallel of testing with Access and Reference HIV Ag/Ab combo assays
  Groups: Known Acute HIV-1 p24 Ag positive
Diagnostic Test: Access HIV_Canada's requirements_Blood donor — To fit with Canada's requirements:
  * 4,000 additional blood donor samples from geographically distinct regions will be collected and tested. Blood donor sample testing will be equally distributed over three blood donor sites, using 3 different lots of reagents: the first 2,000 blood donor samples from CE-marking study (out of the 6,000 tested) will be used plus the 4,000 additional blood donor samples.
  * Retesting of 1000 blood donor samples will be done internally with 1 lot close to expiration to satisfy Canadian requirements
  Groups: Unselected blood donors
Diagnostic Test: Access HIV_Canada's requirements_HIV positive — To fit with Canada's requirements:
  o HIV positive samples will be equally distributed and tested at leat three (3) testing sites, using 3 lots of reagents.
  Groups: Known Acute HIV-1 p24 Ag positive; Known HIV-1 Ab positive; Known HIV-2 Ab positive
Diagnostic Test: Access HIV_Canada's requirements_P24 Positive — To fit with Canada's requirements:
  * HIV positive samples will be equally distributed and tested at leat three (3) testing sites, using 3 lots of reagents.
  * Collection and testing of maximum 210 additional HIV-1 Ag positive sample beyond the 50 required by CTS
  Groups: Known Acute HIV-1 p24 Ag positive

SUMMARY:
The objective of this study is the collection and testing of clinical samples to determine the clinical performance of the Access HIV Ag/Ab Combo assay on the DxI 9000 Access Immunoassay Analyzer

DETAILED DESCRIPTION:
The study will involve a multicenter, prospective and retrospective sample collection, and testing of samples with the investigational HIV assay as required per the EU Common Technical Specification (CTS). The CTS requires testing of samples from blood donors, hospitalized patients, known HIV-1 Ab positive patients, known HIV-2 Ab positive patients, and known HIV-1 p24 Ag positive patients. Any retrospectively collected samples will meet all inclusion/exclusion criteria.

All samples collected will be anonymized or pseudo-anonymized, leftover, remnant samples. pseudo-anonymized collection of samples will required oral patient consent documented in their medical record or electronic case report form (eCRF). For CE marking, below is the number of samples that will be included per group :

* Unselected blood donors : 6,000 fresh samples (requirements CTS : 5,000)
* Hospitalized patients : 1,200 frozen samples and 800 fresh samples (requirements CTS : 200)
* Known HIV-1 Ab positive : 470 frozen samples and 30 fresh samples (requirements CTS : 400)
* Known HIV-2 Ab positive : 100 frozen samples (requirements CTS : 100)
* Known acute HIV-1 p24 Ag positive : 50 frozen samples (requirements CTS : 50)

The following additional design requirements will be incorporated to EU study to satisfy Canadian regulations, but additional data generated on the additional samples will not be used for CE-marking:

* Collection and testing of 4,000 additional blood donor samples. Blood donors' samples should include 300 blood donor matched fresh plasma and serum samples
* Distribution of blood donor sample testing equally over three (3) blood donor sites, using 3 different lots of reagents
* Retesting of 1000 blood donor samples internally with 1 lot close to expiration
* Collection and testing of maximum 210 additional p24 Ag positive sample beyond the 50 required by CTS
* Distribution of p24 Ag and HIV-1 Ab positive sample testing equally over three (3) testing sites, using 3 different lots of reagents.

Additional Canadian requirements will be covered by US protocol(s) and Verification and validation protocols.

ELIGIBILITY:
Inclusion Criteria:

Anonymized or pseudo-anonymized leftover samples from

* Males or females
* Aged ≥18 years of age
* Belonging to one of the following enrollment groups:

  * Unselected blood donor
  * Hospitalized patient
  * Known HIV-1 antibody positive patients

    * confirmed positive by Immunoblot, Western blot or HIV-1/HIV-2 antibody differentiation test either at time of enrollment vai same study draw or historically from medical record
  * Known HIV-2 antibody positive patients

    * confirmed HIV-2 positive by BioPlex 2200 HIV Ag-Ab Assay
  * Known HIV-1 Ag positive patients

    * For samples from HIV seroconversion panels

      * Tested during EU HIV clinical trial: confirmed positive by screening HIV Ag/Ab combo positive for p24 Ag, and p24 Ag screening test positive (result from CoA or additional testing)
      * Tested as part of seroconversion panel studies (V&V studies): First sample of the panel that is ARCHITECT Ag/Ab combo assay positive or BioPlex 2200 HIV Ag-Ab Assay p24 positive, and p24 Ag test positive (result from CoA or additional R&D testing)
    * For routine clinical samples:

      * Confirmed positive by screening HIV Ag/Ab combo assay positive for p24 Ag , and p24 Ag test positive by confirmatory test, or
      * Confirmed positive by screening HIV Ag/Ab combo assay HIV positive, and p24 Ag test positive by confirmatory test and PCR HIV POS and IB/WB HIV negative or indetermined.
* with at least 2.0 mL leftover EDTA plasma sample from hospitalized patients OR
* at least 1.5 mL leftover EDTA plasma or serum sample from blood donors or known HIV-1 antibody positive patients, with confirmatory test already done as per inclusion criteria OR
* at least 1.0 mL leftover EDTA plasma or serum sample from known p24 Ag positive patients or known HIV-2 antibody positive patients, with confirmatory test already done as per inclusion criteria

Exclusion Criteria:

* Samples from subjects already included in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The test population includes :
  * 6,000 unselected blood donors sample
  * 2,000 hospitalized patients
  * 500 Known HIV-1 Ab positive
  * 100 Known HIV-2 Ab positive
  * 50 Known acute HIV-1 p24 Ag positive
Sampling Method: Non-Probability Sample
Enrollment: 8650 (Actual)
Dates: Start 2019-12-04 (Actual); Primary Completion 2022-06-22 (Actual); Study Completion 2022-09-23 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity | Baseline
  Sensitivity and specificity relative to the final patient HIV infection status determined from confirmatory testing will be calculated.

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - Etablissement Français du Sang (EFS) Hauts-de-France - Normandie, Bois-Guillaume
  - Eurofins Biomnis, Ivry-sur-Seine
  - Qbd, Efs Hfno, Loos
  - UPR Lille, Établissement français du sang Hauts-de-France - Normandie, Loos
  - Laboratoire de Virologie, Laboratoire associé au CNR du VIH, Rouen
  - Cerba Xpert, Saint-Ouen-l'Aumône

IPD SHARING:
Plan to Share IPD: No